CLINICAL TRIAL: NCT05417984
Title: Migration of the Restoris MultiCompartmental Knee Implant System in Robotic-assisted Unicompartmental Kneearthroplasty: a 5 Year Follow up RSA Study
Brief Title: RSA Restoris MultiCompartmental Knee
Status: Not yet recruiting | Type: Observational
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: NL79250.058.21
Record Dates: First submitted 2022-05-30; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Unicompartimental knee arthroplasty; Robotic-assisted knee replacement; Migration
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Restoris MCK — During this study the Restoris MCK will be placed using robotic-assisted surgery. At the time of surgery tantalum markers will be placed in the tibia and femur. With these markers migration of the prothesis can be measured over time using RSA radiographs.

SUMMARY:
Patients with isolated medial compartment arthritis of the knee are commonly treated with unicompartmental knee arthroplasty (UKA). In contrast with total knee arthroplasty (TKA), UKA shows a higher revision rate, which might be due to implant malpositioning and postoperative malalignment of the lower limb and incorrect soft tissue balancing. Nowadays, robotic-assisted UKA is used which improves accurate positioning, optimizes soft-tissue balancing and optimizes radiographic alignment of the implant. The potential benefit could be that this better alignment and positioning results in improved functional outcome and long-term survivorship. As there is a lack in long-term results, more research is needed to the long-term results of robotic-assisted UKA. As long-term results are related to early migration of the implant, investigating the early migration will have additional value to predict the long-term results of robotic-assisted UKA. In this study, we will investigate the early migration of a unicompartmental knee implant (Restoris MultiCompartmental Knee Implant System (Restoris MCK)) used in robotic-assisted UKA using model-based roentgen stereogrammetric analysis (mRSA) and we will relate the migration of this implant to the long-term results of the implant.

The primary objective is to assess the fixation and migration patterns of the Restoris MutliCompartmental Knee Implant System (Stryker) in vivo, using mRSA, over 5 years. Secondary objectives are to analyse survival, clinical scores and radiographic aspects of the Restoris MultiCompartmental Knee Implant System (Stryker) and to relate these to the migration patterns over 5 years.

A prospective cohort study with 5 years follow-up, in which 33 patients will be enrolled. Patients 18 years or older who require a unicompartmental knee prosthesis as a result of moderately disabling joint disease of the knee will be included. During surgery tantalum markers will be placed to be able to perform mRSA. Patients will be evaluated preoperatively, at 6 weeks, 6 months, 1 year, 2 years and 5 years.

The main study parameters are the migration of the Restoris MCK of both the tibial and femoral component presented in x-, y- and z-direction. Secondary study parameters are the alignment, survival of the Restoris MCK, clinical scores and radiographic aspects (both x-ray and CT scan).

ELIGIBILITY:
Inclusion Criteria:

* Indication for medial unicompartmental knee replacement as described in the manufacturer's guideline, namely as a result of moderately disabling joint disease of the knee resulting from:

  * Painful osteo- or post-traumatic arthritis
  * As an alternative to tibial osteotomy
* Age > 18 years
* Patient qualified for UKP based on physical exam and medical history
* Patient is able to speak and write Dutch
* Patient is willing to participate
* Patient is able and willing to provide written informed consent

Exclusion Criteria:

* Contraindication as described by the manufacturer:

  * Inflammatory arthritis or tricompartmental disease
  * Greater than 10 degrees of hyperextension
  * Greater than 10 degrees of varus or valgus deformity
  * Presence of infection (including history of infection), acute or chronic, local or systematic
  * Either mental or neuromuscular disorders that do not allow control of the knee joint
  * Insufficient bone stock to allow appropriate insertion and fixation of the prosthesis
  * Insufficient soft tissue integrity to provide adequate stability
  * Insufficient articulation of the hip joint
* Metal in the operative or non-operative leg which lead to the creation of accuracy-reducing artefacts in the CT scan
* Insufficient bone quality to provide adequate stability
* Loss of ligament structures to prevent creation of an ideal intra-operative plan
* Patients has a known or suspected sensitivity or allergy to one or more of the implant materials
* Revision UKP surgery of the same compartment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of all patients who present at the Reinier Haga Orthopedisch Centrum, require unicompartmental knee prosthesis (UKP) and satisfy the inclusion and exclusion criteria as stated below.
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Translation along x-, y- and z-axes | 5 years after surgery at the following time points: 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The translation of both the tibial and femoral component is expressed in mm and is given in 3 directions, namely along the x-, y- and z-axes.
Rotation about x-, y- and z-axes | 5 years after surgery at the following time points: 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The rotation of both the tibial and femoral component is expressed in degrees and is given in 3 directions, namely about the x-, y- and z-axes.

SECONDARY OUTCOMES:
Survival | 5 years after surgery
  Survival of the Restoris MCK is measured by registration of all complications and is expressed by numbers and percentages.
NRS Pain | 5 years after surgery at the following time points: preoperative, 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The Numeric Pain Rating Scale (NRS) measures the amount of pain experienced in the past week during rest and activity. It is a scale from 0 (no pain) to 10 (worst pain imaginable).
KSS | 5 years after surgery at the following time points: preoperative, 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The Knee Society Score (KSS) is a questionnaire to rate the knee prosthesis function. A high score means a good function and a low score means a worse function. The score varies between 0 and 100.
ROM | 5 years after surgery at the following time points: preoperative, 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The Range of Motion (ROM) will be measured during the visit. ROM is the capability of a joint to go through its complete spectrum of movements and is expressed in degrees.
KOOS-PS | 5 years after surgery at the following time points: preoperative, 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The Knee Injury and Osteoarthritis Outcome Score - short version (KOOS-PS) is a questionnaire about the ability to perform normal daily activities. A high score means that the activities cost a lot of effort to perform, while a low score means that the activities can be done with minimum effort. The score varies between 0 and 100.
OKS | 5 years after surgery at the following time points: preoperative, 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The Oxford Knee Score (OKS) is a questionnaire about the amount of influence of the operated knee on the persons life. A low score means that the life of the person is influenced a lot by the operated knee, while a high score means that the life of the persons is little influenced by the operated knee. The score varies between 0 and 48.
EQ-5D-5L | 5 years after surgery at the following time points: preoperative, 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The EuroQol-5D-5L (EQ-5D-5L) is a questionnaire that describes the overall health condition of the person. The score is given by an index consisting of 5 numbers, which reprensents a health status.
FJS | 5 years after surgery at the following time points: 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The Forgotten Joint score (FJS) is a questionnaire about the awareness of the prosthetic knee. A high score means a low awareness and a low score means a high awareness. The score varies between 0 and 100.
Satisfaction | 5 years after surgery at the following time points: 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  The satisfaction is a single question about the overall satisfaction of the result of the surgery on a scale from 0 (very unsatisfied) to 10 (very satisfied).
Radiographic aspects | 5 years after surgery at the following time points: preoperative, 6 weeks, 6 months, 1 year, 2 years and 5 years postoperative.
  Radiographic aspects will be reported and will be described in numbers with percentages.

IPD SHARING:
Plan to Share IPD: Undecided